CLINICAL TRIAL: NCT01450969
Title: Prospective Randomized Evaluation of a New Fabric Attenuation Device in Endovascular Interventional Radiology (PREFER)
Brief Title: New Fabric Attenuation Device in Endovascular Interventional Radiology (PREFER)
Acronym: PREFER
Status: Completed | Type: Observational
Sponsor: Baptist Health South Florida (Other)
Responsible Party: Principal Investigator, Raul Herrera, MD, Director, Division of Clinical Research & Outcomes, Baptist Health South Florida
Other Study IDs: 11-052
Record Dates: First submitted 2011-09-28; First posted 2011-10-13 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Exposure
Keywords: Operator Comfort Assessment; Radiation protection; Measurement of Radiation Exposure; Endovascular Interventional Radiology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Interventional Radiologists: All operators are Interventional Radiologists and co-investigators. Prior to start of the study, all operators are asked to provide written informed consent to participate in the study.

SUMMARY:
The PREFER Trial primary objective of the trial is to show how much radiation attenuation is provided by XPF in absolute and relative terms.

DETAILED DESCRIPTION:
The PREFER Trial has three main objectives. The primary objective of the trial is to show how much radiation attenuation is provided by XPF in absolute and relative terms. The secondary objective of the study is to measure and compare the amount of radiation that interventional radiologists are exposed to per case in an interventional suite setting using FDA approved XPF thyroid collars or standard 0.5 mm Pb equivalent thyroid collars. The third objective is to assess the operator comfort wearing the XPF protection devices. In order to achieve these objectives, measurements will be performed in 60 consecutive endovascular procedures requiring C-arm fluoroscopy performed at BCVI. Participants will be asked to wear an XPF cap (weighing approximately 100 grams) in every study procedure. Furthermore, a prospective randomization will be performed, assigning participants to wear their own standard 0.5 mm Pb equivalent thyroid collar or to wear the FDA approved XPF thyroid collar. Radiation exposure will be monitored with 4 radiation detectors (TLDs, 2 attached to the cap, 2 attached to the collar) which the participant is required to wear. After each procedure the participant will be asked to rate the comfort of wearing the devices on a scale from 1 to 100.

ELIGIBILITY:
Inclusion Criteria:

* Interventional Radiologists practicing in Baptist Cardiac & Vascular Institute
* consecutive endovascular procedure requiring C-arm fluoroscopy

Exclusion Criteria:

* Interventional Neuroradiologists and Interventional Cardiologists will not be included in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All operators are Interventional Radiologists and Co-Investigators. Prior to start of the study, all operators are asked to provide written informed consent to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-09; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Radiation attenuation in percentage (%) and in absolute terms (μSv/min) | The attenuation is assessed directly after each procedure (day 1)
  The null hypothesis is that the XPF thyroid collar is inferior to the standard 0.5mm Pb lead equivalent thyroid collar with regard to radiation attenuation/transmission. The alternative hypothesis is that the XPF thyroid collar is non-inferior to the standard thyroid collar. If there is truly no difference between standard and XPF thyroid collars, then 60 patients are required to be 95% sure that the lower limit of a one-sided 95% confidence interval (or equivalently a 90% two-sided confidence interval) will be above the non-inferiority limit of -0.7% transmission rate and -0.013 μSv/min.

SECONDARY OUTCOMES:
Wearing comfort of the XPF cap and collar on a scale from 0-100. | (day 1) Operators are asked directly after each procedure to rate the wearing comfort

CONTACTS AND LOCATIONS:
Overall Officials: Barry T. Katzen, MD, Principal Investigator — Baptist Hospital of Miami and its Miami Cardiac and Vascular Institute; Heiko Uthoff, MD, Principal Investigator — Baptist Hospital of Miami and its Miami Cardiac and Vascular Institute
Locations (1):
- Baptist Hospital of Miami, Miami Cardiac and Vascular Institute, Miami, Florida, United States